CLINICAL TRIAL: NCT01349582
Title: A Randomized Trial Comparing Flow Diversion and Best-standard Treatment - the FIAT Trial
Brief Title: Flow Diversion in Intracranial Aneurysm Treatment
Acronym: FIAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE10.206
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Intracranial Aneurysm
Keywords: flow diversion; endovascular treatment; symptomatic aneurysm; cavernous carotid aneurysm; ophthalmic aneurysm; vertebral aneurysm
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- flow diversion (Active Comparator): Flow diverters are low porosity braided endovascular stent devices. They can be used with or without coiling.
  Interventions: Procedure: flow diversion
- Best standard treatment (Active Comparator): Best standard treatment can by any of the standard management options: coiling, stenting plus coiling, surgical clipping, parent vessel occlusion, observation
  Interventions: Other: conservative management; Procedure: endovascular coiling; Procedure: balloon parent vessel occlusion; Procedure: surgical clipping
- Registry for flow diversion (Other): Flow diversion when randomization between flow diversion and best standard treatment is not possible and the only alternative is flow diversion for compassionate use. In this case there will be no random allocation but the patient will be entered into a registry
  Interventions: Procedure: flow diversion

INTERVENTIONS:
Procedure: flow diversion — endovascular treatment with flow diversion including standard management of thrombo-embolic risk
  Arms: Registry for flow diversion; flow diversion
Other: conservative management — conservative management is watchful observation of the aneurysm until indication for intervention arises
  Arms: Best standard treatment
Procedure: endovascular coiling — standard endovascular coiling of aneurysm with any type of already approved coil. High porosity stents may be used as an adjunct technique to coiling
  Arms: Best standard treatment
Procedure: balloon parent vessel occlusion — sacrifice of parent artery of aneurysm by endovascular balloon occlusion with or without bypass
  Arms: Best standard treatment
Procedure: surgical clipping — clipping of the aneurysm following invasive brain surgery
  Arms: Best standard treatment

SUMMARY:
Flow diverters are a recent addition to the range of endovascular devices now available for the treatment of intracranial aneurysms. The FIAT trial aims at comparing flow diversion to best standard treatment in the context of a randomised controlled trial. Best standard treatment may include any of the following and will be left to the treating physician to decide : 1) conservative management; 2) coiling with or without high porosity stenting; 3) parent vessel occlusion with or without bypass; 4) surgical clipping. If the only treatment alternative is deemed to be flow diversion for compassionate use, then randomisation will not be carried out, but patient will enter a registry and her data recorded according to same schedule as randomised patients.

The primary hypothesis is that flow diversion can be performed with an "acceptable" immediate complication rate, defined as less than 15% morbidity and mortality, AND increase the number of patients experiencing successful therapy, defined as complete or near complete occlusion of the aneurysm from 75 to 90%, relative to best standard treatment.

DETAILED DESCRIPTION:
Background:

Intracranial aneurysms, particularly large/giant, fusiform or recurrent aneurysms are increasingly treated with flow diverters (FDs), a recently introduced and approved neurovascular device. While some rare cases may not be treated any other way, in most patients a more conventional, conservative, or validated approach such as coiling, parent vessel occlusion, or surgical clipping exists. Early series and registries of the use of FDs in various types of aneurysms have reported treatment-related morbidity and mortality ranging from 0 to 4 and 8% respectively, most often from delayed haemorrhage. Hence, although there is growing enthusiasm to use these powerful new tools, complications are increasingly reported.

Rationale and Hypothesis:

There is an urgent need to offer the new tool afforded by FDs to patients currently presenting with a difficult aneurysm, in a context that can offer protection from over-optimistic perspectives, fashion, learning curves and marketing. Only a randomized clinical trial can offer such protection as well as provide an answer to the question of which treatment option leads to better patient outcomes. The primary hypothesis is that flow diversion can be performed with an "acceptable" immediate complication rate, defined as less than 15% morbidity and mortality (modified Rankin Score > 2 at 3 months), AND increase the number of patients experiencing successful therapy, defined as complete or near complete occlusion of the aneurysm from 75 to 90%.

Objectives:

Compare flow diversion (FD) to Best-Standard Treatment (BST) in the context of an RCT. BST may be any of the following: 1) conservative management; 2) coiling with or without high porosity stenting; 3) parent vessel occlusion with or without bypass; 4) surgical clipping; 5) enter a registry for FD, when the only treatment alternative is FD for compassionate use.

Methods:

Following randomization to FD or BST, patients will undergo the assigned intervention and be followed for 12 months. Clinical status will be recorded at discharge, at 1-3 months, and at 3-12 months. Angiographic evaluation will be recorded at 3-12 months. Adverse Events will be recorded immediately after the procedure and during the 12-month follow-up period. Patients in the FD registry will similarly be followed for 12 months. A total of 344 patients will be recruited in 20 centers worldwide. The trial is expected to last for 5 years.

Analysis:

Comparability between FD and BST groups will use descriptive statistics or frequency tables, independent ANOVAs or Mantel-Haentzel and chi-square tests. Comparison of primary outcome will use a z-test for independent proportions at 12 months. Safety data will be compared through independent t-tests or chi-square statistics. Logistic regression will be used to find variables capable of predicting success in both groups at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a "difficult" intracranial aneurysm in whom flow diversion is considered an appropriate if not the best but yet unproved therapeutic option by the participating clinician. Current indications may be (but not restricted to) symptomatic large or giant cavernous carotid, ophthalmic and vertebral aneurysms, fusiform intradural aneurysms, or recurring, persistent lesions after previous coiling. Aneurysm may be a recent rupture, although risks associated with antiplatelet regimens in this context should make this option rarely used

Exclusion Criteria:

* Severe allergy, intolerance or bleeding disorder that prohibit the use of ASA or clopidogrel.
* Absolute contraindication to endovascular treatment or anesthesia.
* Patients unable to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2011-05-02 (Actual); Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
rate of success of therapy | 12 months
  Rate of success increases from 75% to 90%, with success defined as complete or near complete occlusion of the aneurysm combined with a modified Rankin score of less or equal to 2.

SECONDARY OUTCOMES:
modified Rankin score | discharge, 3 and 12 months
  modified Rankin score at discharge, and at 3 and 12 months post-treatment (last observation carried forward)
rate of peri-operative complications | 30 days
  rate of ischemic strokes and intracranial hemorrhages during the peri-operative period
rate of Adverse Events | 12 months
  rate of new stroke, neurological symptom or sign during follow-up
angiographic outcome | 12 months
  degree of occlusion of aneurysm as assessed by invasive or non-invasive imaging (last observation carried forward
rate of retreatment of index aneurysm | 12 months
  rate of retreatment of index aneurysm due residual aneurysm after initial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean Raymond, MD, Principal Investigator — Centre Hospitalier de l'Université de Montréal - Hôpital Notre Dame
Locations (3):
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - The Ottawa Hospital, Ottawa, Ontario
  - Centre Hospitalier de l'Université de Montréal - Hôpital Notre Dame, Montreal, Quebec

REFERENCES:
- [Derived] Raymond J, Gentric JC, Darsaut TE, Iancu D, Chagnon M, Weill A, Roy D. Flow diversion in the treatment of aneurysms: a randomized care trial and registry. J Neurosurg. 2017 Sep;127(3):454-462. doi: 10.3171/2016.4.JNS152662. Epub 2016 Nov 4. PMID 27813466